CLINICAL TRIAL: NCT02311192
Title: Grading Scale of Vitreous Haze in Patients With Uveitis Using Ultrasonography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Department chair choose not to participate
Sponsor: University of Nebraska (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Luigi Sacco University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0583-14-EP
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Uveitis
Keywords: Vitreous Haze; Ocular ultrasound; B scan; Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ultrasonography B-scan (Experimental): Patients of uveitis who are included in the study will be imaged using ultrasound B-scan
  Interventions: Device: Ultrasonography B-scan

INTERVENTIONS:
Device: Ultrasonography B-scan — The patient's eye will be anesthetized. The ultrasound probe will then be used to obtain images by keeping the probe in light contact with the eye.

SUMMARY:
This study is aimed at creation and validation of a vitreous haze scoring system using ultrasonography B-scan of the eye. Images will be obtained from patients with uveitis and quantification of inflammation will be done to create the scoring scale.

DETAILED DESCRIPTION:
Patients with uveitis may present with Vitreous Haze (VH) resulting in obscuration of fundus details. VH is composed of cells and protein exudation and results in decrease visual acuity.The degree of VH is an important indicator of disease activity, severity and response to therapy in patients with uveitis. Color fundus images are commonly used to objectively document VH.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to provide written informed consent and comply with study assessments for the full duration of the study

  * Age 18 -90 years
  * Diagnosis of uveitis

Exclusion Criteria:

* • Patients with posterior segment complications including retinal detachment, choroidal detachment or hemorrhage

  * Patients with any intraocular foreign body or displaced intraocular lens
  * Patients with silicon oil filled eye or with gas tamponade.
  * Patients with vitreous hemorrhage
  * Patients with media opacity including visually significant cataract that precludes grading of VH based on fundus photography

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Inter-observer correlation for vitreous haze grading | 1 year
  Inter-observer correlation for vitreous haze (VH) grading will be assessed using number of eyes as the unit of measure as well as standardized grading scheme for VH

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD MSc, Principal Investigator — University of Nebraska; Giovanni Staurenghi, MD, Principal Investigator — Luigi Sacco Hospital; Ramandeep Singh, MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh